CLINICAL TRIAL: NCT04775134
Title: Residual SARS-CoV-2 Presence in the Respiratory Tract and Lung Parenchyma
Brief Title: Residual SARS-CoV-2 Presence in the Respiratory Tract and Lung Parenchyma (After SARS-CoV-2 Infection or COVID-19)
Acronym: REASSURE
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64988
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects with earlier PCR-proven COVID-19 and/or serum anti-SARS-CoV-2 antibodies: Patients that require a medically indicated pulmonary resection.
  Interventions: Diagnostic Test: Lung biopsy
- Subjects WITHOUT earlier PCR-proven COVID-19 and/or serum anti-SARS-CoV-2 antibodies: Patients that require a medically indicated pulmonary resection.
  Interventions: Diagnostic Test: Lung biopsy

INTERVENTIONS:
Diagnostic Test: Lung biopsy — Biopsy of residuary material from a medically indicated pulmonary resection

SUMMARY:
The aim of this study is to confirm or rule out the residual presence and viability of SARS- CoV-2 in the respiratory tract and lung parenchyma of patients previously infected with SARS-CoV-2.

Presence and viability of SARS-CoV-2 in lung tissue will be assessed with reverse transcriptase-polymerase chain reaction (PCR) and viral culture. The histological location of residual SARS-CoV-2 will be determined with fluorescence immunohistochemistry and single molecule fluorescence in situ hybridization, targeting viral proteins and RNA respectively.

DETAILED DESCRIPTION:
The investigators will collect residuary lung tissue after medically indicated pulmonary resections at the Thoracic Surgery Department of University Hospitals Leuven. More specifically the investigators will collect lung tissue from patients that had earlier PCR proven COVID-19 and/or serum anti-SARS-CoV-2 antibodies.

Furthermore, for negative control of the methodology the investigators will also collect lung tissue from patients that have no signs for earlier SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires medically indicated pulmonary resection
* Informed consent

Exclusion Criteria:

* Active SARS-CoV-2 infection/COVID-19
* No informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients requiring a medically indicated pulmonary resection.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reverse transcriptase-PCR | Single time point.
  Detection of SARS-CoV-2 RNA in lung tissue homogenate with primers targeting both genomic and subgenomic RNA
Fluorescence immunohistochemistry (IHC) | Single time point.
  Determining the histological presence of SARS-CoV-2 viral proteins in lung tissue with commercially available antibodies against the SARS-CoV-2 spike and nucleocapsid proteins
Single molecule fluorescence in situ hybridization (smFISH) | Single time point.
  Determining the presence of SARS-COV-2 viral RNA in lung tissue with commercially available probes targeting both sense and anti-sense viral RNA

SECONDARY OUTCOMES:
Viral culture | Single time point.
  Determining viability of SARS-CoV-2 in case of a low revere transcriptase-PCR cycling threshold

CONTACTS AND LOCATIONS:
Overall Officials: Laurens J Ceulemans, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided